CLINICAL TRIAL: NCT03490786
Title: A Dose Escalating Study to Assess the Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of a Lingual Application of GT-001 in Subjects With Obesity.
Brief Title: A Dose Escalating Study to Assess the Safety and Tolerability of GT-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gila Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2018-02-19; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Feeding and Eating Disorders
Keywords: GT-001
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — peptide YY (3-36)

STUDY DESIGN:
Intervention Model Description: dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): Single arm dose escalation.
  Interventions: Drug: GT-001

INTERVENTIONS:
Drug: GT-001 — PK, PD Study to Determine Safety of Escalating Doses of GT-001
  Other Names: PYY(3-36); Peptide YY (3-36)

SUMMARY:
Dose escalation study of GT-001

DETAILED DESCRIPTION:
This is a dose-escalation design trial. Twelve evaluable subjects (n=12) with BMIs of 30 to 40 kg/m2 will receive a single dose of placebo followed by study drug applied directly to the surface of the tongue mucosa with a disposable pipette followed by a one-day washout. A total of seven (7) doses will escalate to a dose of 2.5 mg.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with obesity class I and II (BMI 30-40 kg/m2)
* Willing and able to provide written informed consent after reviewing the design and risks of the study and prior to completing any study-related procedure
* Willing and able to understand and comply with all study procedures and requirements.
* Women must have a predictable menstrual cycle and taking either monophasic oral contraceptives, or transdermal (Ortho Evra and Evra) at least one month prior to the study.
* Alternatively, post-menopausal women (defined as period of spontaneous amenorrhea for more than 1 year), and bilateral oophorectomized women are allowed into the study.
* Must be able to complete the Weight Efficacy Life-Style Questionnaire (WEL).
* Systolic blood pressure 100-160 mmHg at the time of screening.
* Stable and compliant treatment with oral medications for at least 4 weeks prior to screening.
* Women of child bearing potential (WOCBP) and males must agree to use at least two forms of contraception, of which one includes a barrier method (male condom) by the male partner, during study participation and continued for at least 90 days after the conclusion of the final dose.
* In addition, sperm donations by male subjects are not permitted during the subject's participation in the research study and for at least 90 days after the conclusion of the final dose. This criterion may be waived for male subjects who have undergone a vasectomy at least 6 months prior to screening.
* Willing and able to abstain from drugs, , and tobacco during study participation.
* Must have abstained from alcohol use for 48 hours prior to study day 1 through the duration of the study
* Must have abstained from any tobacco- or nicotine-containing products (e.g., cigarettes, e-cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to study day 1.
* History of stable weight for at least 3 months prior to study entry.

Exclusion Criteria:

* Known hypersensitivity or allergy to Peptide YY, Pancreatic polypeptide (PP), other similar polypeptides or related compounds
* Known mutation to PYY or Y2 receptor gene (i.e., Pima Indians)
* Any medical condition for which modification of the medication that cannot be performed either safely or feasibly. Chronic diseases including metabolic, psychiatric, cardiovascular, endocrine, etc. for which the participant is not stable for 60 days prior to study initiation
* Female subjects who are pregnant or breast-feeding
* Female subjects of child bearing potential who are not on oral contraceptives or using biphasic or triphasic oral contraceptives
* Post-menopausal women who have not had a period of spontaneous amenorrhea for more than 1 year Unstable psychological or behavior profile (e.g., anxiety, depression)
* Subjects with fasting glucose levels greater than 125 mg/dl.
* Type I or Type II diabetes
* Poor dentition or oral pathology
* Unable or unwilling to give written informed consent.
* Temperature > 38°C (oral or equivalent)
* Sepsis or active infection requiring IV antimicrobial treatment
* Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (not including restrictive mitral filling patterns)
* Major neurologic event, including cerebrovascular events within 60 days prior to study initiation
* Significant pulmonary disease (e.g., history of oral daily steroid dependency, history of CO2 retention or need for intubation for acute exacerbation, or currently receiving IV steroids)
* Known hepatic impairment as indicated by any of the following:

  * Total bilirubin > 3 mg/dl
  * Albumin < 2.8 mg/dl, with other signs or symptoms of hepatic dysfunction
  * Increased ammonia levels, if performed, with other signs or symptoms of hepatic dysfunction
* Any organ transplant recipient or currently listed (anticipated in the next 60 days) for transplant
* Major surgery within 30 days prior to study initiation
* Positive screen for Hepatitis B (HbsAg, Hepatitis B Surface Antigen), Hepatitis C (anti-HCV, Hepatitis C Antibody), or HIV (anti-HIV 1/2)
* Received an investigational intervention within 30 days prior to study initiation, or have received PYY3-36, GLP-1 agonists, insulin or DPP-IV inhibitors in a previous clinical trial.
* Consumption of alcohol within 48 hours prior to study day1 and through study day 15 or early termination
* Use of any tobacco- or nicotine-containing products (e.g., cigarettes, e-cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months
* A positive urine drug screen for ethanol, cotinine, cocaine, THC, barbiturates, amphetamines, benzodiazepines, and/or opiates
* A history of difficulty with donating blood, or having donated blood or blood products within 45 days prior to study initiation
* Use of weight loss drugs Orlistat (Alli or Xenical), Qsymia, Phentermine, Contrave, Lorcaserin, liraglutide, topiramate or exenatide within the last six months.
* Concurrent use of antihistamines
* Any condition that, in the opinion of the Investigator or Medical Monitor, would render the subject unsuitable for participation in the study
* Unable to consume the test meal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-16 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Demonstrate safe doses of PGT-001 for reduction of body weight in obese volunteers. | approximately two weeks
  Measures of the safety and tolerability of GT-001 include documentation of adverse events and changes (compared to baseline) in vital signs, physical examination, and laboratory tests.

SECONDARY OUTCOMES:
Dose-relationship of adverse events | approximately two weeks
  Incidence, severity and dose-relationship of adverse events as well as changes in physical examinations, vital signs and/or laboratory evaluations as a measure of safety and tolerability.
Dose relationship to peak plasma concentration of GT-001 | Approximately two weeks
  Peak plasma concentration of GT-001 to assess relationship to dose of GT-001.
Dose relationship to hunger and satiety | approximately two weeks
  Measurement of hunger and satiety will be conducted using visual analog scores to assess a relationship to dose of GT-001

CONTACTS AND LOCATIONS:
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No